CLINICAL TRIAL: NCT01034345
Title: Effect of Rapamycin on Tolerance-related Biomarkers on Stable Liver Transplant Recipients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Alberto Sanchez-Fueyo, Hospital Clinic Barcelona/ IDIBAPS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sirolimus_Liver_Tolerance
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Last update posted 2009-12-17 (Estimated); Status verified 2009-11

CONDITIONS: Liver Transplantation
Keywords: Sirolimus; Liver Transplantation; Tolerance; Immune responses; Allograft tolerance
MeSH Terms: interventions — Sirolimus; Calcineurin Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sirolimus (Experimental): Patients randomized to this arm will discontinue maintenance immunosuppression based on calcineurin inhibitors and start treatment with sirolimus.
  Interventions: Drug: Sirolimus
- Calcineurin inhibitor (Active Comparator): Patients randomized to this arm will keep the same maintenance immunosuppression based on calcineurin inhibitors.
  Interventions: Drug: Calcineurin inhibitor

INTERVENTIONS:
Drug: Sirolimus — Switch from calcineurin inhibitor maintenance immunosuppression to sirolimus treatment at the doses needed to reach trough blood levels 8-15 ng/mL.
  Arms: Sirolimus
Drug: Calcineurin inhibitor — Patients will maintain the same immunosuppressive regimen based on calcineurin inhibitors. No modifications in the treatment will be conducted.
  Arms: Calcineurin inhibitor

SUMMARY:
In contrast to calcineurin inhibitors, sirolimus is known to exert remarkable tolerance-promoting properties in multiple animal transplant models. Whether sirolimus is capable of enhancing tolerance-related pathways and/or promoting complete withdrawal of immunosuppressive drugs in human transplant recipients has not been previously addressed. The goal of the investigators study is to evaluate the effects of sirolimus on previously identified tolerogenic pathways in humans and, indirectly, to assess the capacity of this drug to enhance the proportion of liver recipients undergoing successful immunosuppression weaning.

DETAILED DESCRIPTION:
Objective:To test in liver transplant recipients identified as non-tolerant whether discontinuation of calcineurin inhibitors followed by 6-month treatment with sirolimus modifies the pattern of expression of the set of genes associated with tolerance

Background: Sirolimus is an immunosuppressive drug used to counter autoimmunity and to prevent acute graft rejection in human and has remarkable tolerance-promoting properties in animal transplant models.

Hypothesis/Specific Aims:We hypothesize that sirolimus promotes tolerogenic pathways in human liver transplantation.

1. To test in liver transplant recipients identified as non-tolerant whether discontinuation of calcineurin inhibitors followed by 6-month treatment with sirolimus modifies the pattern of expression of the set of genes associated with tolerance
2. To test in liver transplant recipients identified as non-tolerant whether conversion from calcineurin inhibitors to sirolimus modifies memory type immune responses.
3. To test in liver transplant recipients identified as non-tolerant whether conversion from calcineurin inhibitor monotherapy to sirolimus affects the frequency, phenotype and function of potentially immunoregulatory peripheral blood lymphocyte subsets
4. To test in liver transplant recipients identified as non-tolerant whether conversion from calcineurin inhibitors to sirolimus promotes epigenetic changes related to immunoregulation and cancer development/progression

Proposed Methods:Gene expression experiments: we will quantify the expression in peripheral blood of a set of genes previously identified as predictive of successful immunosuppression withdrawal in stable liver transplant recipients. Blood samples will be obtained before and 6 months after conversion to sirolimus treatment. Measurement of gene expression levels will be conducted employing real-time TaqMan PCR. Classification of patients in the tolerant/non-tolerant categories will be conducted utilizing thresholds and predictive algorithms developed in our laboratory.

Immunophenotyping studies: we will quantify in peripheral blood various mononuclear cell subsets implicated in immunoregulatory pathways before and 6 months after conversion to sirolimus treatment. Measurements will be conducted employing flow cytometry.

Functional assays: we will isolate CD4+CD25+ regulatory T cells (Treg) from peripheral blood by Sorter before and 6 months after conversion to sirolimus treatment. Serial dilution experiments will be conduct in an antigen non-specific assay to assess the relative suppressive properties of Tregs. IFNg ELISpot assays will be conducted in parallel employing peripheral blood mononuclear cells as responder cells to measure donor-specific alloimmune responses.

Measurement of DNA-methylation: recipient DNA will be extracted from peripheral blood samples before and after 6-month sirolimus treatment and used to conduct whole-genome methylation studies employing the ILLUMINA array platform.

Expected results: We expect to precisely define the effects of sirolimus on previously identified tolerogenic pathways in humans and, to assess the capacity of this drug to enhance the proportion of liver recipients undergoing successful immunosuppression weaning.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and weight ≥ 40 kg
* Women of childbearing potential must have a negative serum pregnancy test result before random assignment and must agree to use a medically acceptable method of contraception throughout the treatment period and for 3 months after discontinuation of randomly assigned treatment. Any woman becoming pregnant during the treatment period must withdraw from the study
* Subjects receiving immunosuppressive therapy with a stable regimen of calcineurin inhibitor or a combination of calcineurin inhibitor with corticosteroids and/or antimetabolite therapy for a minimum of 4 weeks prior to randomization
* Recipient of a liver transplantation with >3 years follow-up Cockcroft-Gault GFR values ≥ 40 mL/min
* Total white blood cell count >3.0 x 109/L (>3,000/mm3), platelet count >75 x109/L (>75,000/mm3), fasting triglycerides <3.95 mmol/L (<350 mg/dL), fasting cholesterol <7.8 mmol/L (<300 mg/dL). If subjects are currently untreated for elevated cholesterol and/or triglycerides and are excluded from the study based on the above criteria, subjects will be offered antihyperlipidemic therapy.
* Stable liver function defined as: a) normal liver function tests (AST, ALT, ALP, GGT) during the previous 6 months; or alternatively b) minor alterations in liver function tests that have not changed over the previous 6 months (AST/ALT < 2 fold normal levels; ALP < 1.5 fold normal levels; GGT < 3 fold normal levels; bilirubin < 3 mg/dL).
* Absence of treatment with interferon for hepatitis C virus infection
* Absence of autoimmune diseases requiring immunosuppressive therapy
* Absence of autoimmune liver disease as indication for transplantation
* Absence of any rejection episodes in the 12 previous months
* Peripheral blood gene expression profile characteristic of non-tolerant recipients (likelihood of successful weaning <5%)
* Written, signed, and dated IRB- or IEC-approved informed consent

Exclusion Criteria:

* Requirement for treatment with immunosuppressive drugs for any indications other than prevention of rejection
* Proteinuria levels > 0.8 g/day
* Evidence of systemic infection (e,g., sepsis, bacteremia, pneumonia, etc.) at time of random assignment.
* History of documented human immunodeficiency virus infection.
* Hypercoagulable states or any history of deep vein thrombosis, HAT, or portal vein thrombosis. (Exception: incidental vascular thrombosis at the time of liver explant, which in the opinion of the investigator, does not place the subject at increased risk of thrombotic events.)
* Transplant of other graft in addition to the liver

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2009-11; Primary Completion 2011-11 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Effects of conversion from calcineurin inhibitors to sirolimus on tolerance-related biomarkers of tolerance in human liver transplant recipients. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Sanchez Fueyo, MD, Principal Investigator — Hospital Clinic Barcelona/IDIBAPS, University of Barcelona
Locations (1):
- Hospital Clinic Barcelona, University of Barcelona, Barcelona, Barcelona, Spain